CLINICAL TRIAL: NCT06862336
Title: Intradialytic Versus Interdialytic Resistance Exercises on Quality of Life in Patients with Chronic Kidney Diseases
Brief Title: Interdialytic Resistance Exercises in with Chronic Kidney Diseases
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira saad mohamed, lecturer of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012/005019
Record Dates: First submitted 2025-03-02; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): twenty-five patients with CKD will receive intra-dialytic combined exercise program for8 weeks(3 sessions/week), with their medical treatment.
  Interventions: Procedure: intra-dialytic exercise program associated with medical treatment
- Group B (Placebo Comparator): twenty-five patients with CKD will receive the inter-dialytic combined exercise program with their medications.
  Interventions: Procedure: inter-dialytic combined exercise program with their medications

INTERVENTIONS:
Procedure: intra-dialytic exercise program associated with medical treatment — * Stretch for pectorals and calf muscles: Two sets - 3 times/ set.
  * Breathing exercises associated with upper limb movement.
  * Resistive exercise for hip abductors, hip flexors, and calf muscles by using theraband.
  * Sit to stand strengthening exercises: -
  Arms: Group A
Procedure: inter-dialytic combined exercise program with their medications — receive the inter-dialytic combined exercise program with their medications. Like the study group except for diaphragmatic breathing instead of breathing with upper limb exercise.
  Arms: Group B

SUMMARY:
Fifty chronic kidney disease patients' ages will range from 40 to 55 years. They will be selected from the dialysis unit. received intra-dialytic combined exercise program for 8 weeks(3 sessions/week), with their medical treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Fifty patients with CKD, are on hemodialysis for longer than threemonths 3 sessions/ week.
2. Theirageswillrangefrom40 to 55yearsold.
3. Their body mass index is more than 18.5 and less than 29.9 %.

3-All patients have hemodynamic stability over the month before beginning the program.

Exclusion Criteria:

* 1. Severe Chest diseases(either obstructive or restrictive). 2. Clinical signs of a severe cardiac event.(eg, severe atherosclerosis, congestive heart failure), 3. Severepsychiatricorcognitiveimpairment,whounabletofollowcomment. 4. Neurological disorders affecting respiratory muscles or any muscular dystrophies(cervical disc or bulge).

  5. Patients with severe self-limiting illness (e.g., cancer). 6. peripheral artery disease in lower extremities. 7. Systolic blood pressure < 180 mmHg, diastolic blood pressure more than 105 mmHg, or heart rate above 120 bpm during dialysis.

  8. Patient with uncontrolled- diabetes.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-03-20 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Measuring quadriceps and cuff muscles power | pre intervention and re assessed after 2 months of treatment
  From sitting or lying positions the normal dialytic positions by handheld dynamometer

SECONDARY OUTCOMES:
Kidney disease quality of life F | pre intervention and re assessed after 2 months of treatment
  Kidney disease quality of life questionnaire KDQoL-SF
chest expansion | pre intervention and re assessed after 2 months of treatment
  From a standing position and comfortable clothes with relaxed shoulders and a straight back, the head will be aligned vertically. Putting the measuring tape around the armpits and closing the ends of the tape measurement not tightly nor loose, asking the patient to take deep breathing.
Six-minute walk test | pre intervention and re assessed after 2 months of treatment
  Subjects will be instructed to walk from one end to the other of a 30-m hallway at their own pace while attempting to cover as much ground as possible in the allotted 6 min

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Egypt